CLINICAL TRIAL: NCT07148817
Title: Impact of Personal Mitigation on Mechanisms Linking Transportation Noise Exposure to Cardiometabolic Disease
Brief Title: Impact of Earplugs on Mechanisms of Noise-Related Cardiovascular Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Michael T. Osborne, Assistant Professor of Medicine and Cardiologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P001821; 25TPA1474746 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-08-18; First posted 2025-08-29 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Cardiometabolic Diseases; Noise Exposure
Keywords: Transportation Noise; Cardiometabolic Diseases; Earplugs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Earplug use (Active Comparator): Individuals assigned to this group will use earplugs to attenuate noise <45 dB during sleep and rest during the 6 month study period
  Interventions: Behavioral: Noise canceling earplugs
- Control (Placebo Comparator): Individuals assigned to this group will not attempt noise mitigation during sleep and rest during the 6 month study period
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Noise canceling earplugs — Modifiable noise cancelling earplugs will be used to attempt to limit individual noise exposure in those with high levels of exposure or high levels of annoyance related to noise
  Arms: Earplug use
Behavioral: Usual care — No behavioral changes to limit noise exposure
  Arms: Control

SUMMARY:
Noise from cars, planes, and trains affects all people and has been associated with heart disease. Almost 30% of Americans are exposed to harmful levels of noise and noise accounts for the loss of more than one million healthy life years per year in Europe. Noise causes stress and may be most dangerous when it happens at night. The mechanisms linking noise to heart disease involve changes in the brain and the "fight or flight" response. These changes lead to inflammation and blood vessel disease. However, there are few laws that restrict noise and it is not addressed in medical care. Further, as cities and industries grow, noise continues to increase. Moreover, noise often occurs in areas that are also exposed to other stressors like high air pollution and low income. Yet, there is little research on noise, and it is not known if lowering noise exposure helps heart health. The investigators will use imaging to test if earplugs that block noise improve stress symptoms and changes in the the brain, blood vessels, and stress pathways that lead to disease. The investigators expect that people who use earplugs will have lower measures of stress and heart disease at follow-up. The study will include 26 people with heart disease risk with high noise exposure or who are annoyed by noise. At the first visit, subjects will have imaging of the brain and blood vessels and will have assessments of stress, inflammation, and the "fight or flight" response. They will be assigned to use earplugs or not after the first visit. After 6 months, imaging and other testing will be repeated. It will help to understand how noise impacts the body and whether the effects can be changed. It may also identify important treatments to prevent heart disease in people exposed to noise. By testing if the adverse effects of noise can be lowered with earplugs, this project supports the AHA's mission to be a force for a world of longer and healthier lives.

DETAILED DESCRIPTION:
Transportation noise is a pervasive exposure in modern life that has been associated with cardiovascular and metabolic disease. Almost 30% of Americans are exposed to harmful levels of noise and noise accounts for the loss of more than one million healthy life years per year in Europe. Noise exposure leads to activation of the stress response and nocturnal exposure may be more dangerous. The pathologic mechanisms linking noise to cardiovascular disease have recently been shown to involve changes in the metabolic activity of stress responsive brain regions (specifically the ratio of activity in the amygdala to that of the cortex or stress-associated neural activity, SNA) and fluorodeoxyglucose positron emission tomography, FDG PET) and autonomic dysfunction. These changes lead to stress hormone release, inflammation, vascular dysfunction, oxidative stress, increased cardiovascular risk factors, and, ultimately, atherosclerosis. However, there are few laws that restrict noise and it is not addressed in routine medical care. Further, as cities and industries grow, noise exposure continues to increase. Moreover, noise exposure often occurs coincidentally with other psychosocial and environmental stressors, such as high air pollution and low income. Yet, there is little research on noise, and it is not known if personal noise mitigation attenuates the stress response and downstream markers of cardiovascular risk. The investigators will leverage will use advanced FDG PET/magnetic resonance imaging to test if noise canceling earplugs improve stress symptoms and reduce SNA, arterial inflammation, and autonomic and inflammatory intermediaries. The study will assess whether earplug use will decrease SNA and arterial inflammation by attenuating autonomic and inflammatory intermediaries. The investigators will recruit 26 people with cardiovascular risk with high noise exposure or annoyance for this pilot study. At baseline, subjects will have FDG PET/MRI of the brain and aorta and will have assessments of stress, inflammation, and autonomic function. They will be randomized to use earplugs or control. After 6 months, the baseline visit will be repeated. This study will clarify how noise impacts the body and whether its adverse effects can be reduced. It may also identify novel treatments to prevent heart disease in people exposed to noise. By testing if the adverse effects of noise can be mitigated with earplugs, this study takes a necessary step towards reducing noise-related cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Describe feeling annoyed by transportation noise exposure or have high residential noise exposure (>45 dBA average over 24 hours) using the United States Department of Transportation Map
* Known stable atherosclerosis or at least one typical risk factor (i.e., hypertension, diabetes, active smoking, or hyperlipidemia)
* Ability to understand and sign informed consent

Exclusion Criteria:

* History of stroke, brain surgery, or seizure
* Use of certain CVD medications (e.g., beta-blockers, high-intensity statins [e.g., rosuvastatin 20/40 mg and atorvastatin 40/80 mg], PCSK-9 inhibitors)
* Psychiatric or cardiovascular medication change within 3 months (i.e., stable regimen is allowed)
* Unstable blood pressure or cardiac arrhythmia
* Current use of personal noise mitigation techniques or involvement in stress management program
* Moderate/severe alcohol/substance use disorder
* Current mania/psychosis
* Weight >300 lbs.
* Claustrophobia
* Pregnancy
* Metal implants
* Uncontrolled hyperglycemia (HgbA1c>7.5%)
* Subjects who have had significant radiation exposure as part of research (>2 nuclear tests, computed tomography images, or fluoroscopic procedures) during the preceding 12-months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Stress-Associated Neural Activity | Baseline and 6 months
  Measured on FDG-PET as the ratio of metabolic activity of the amygdala to that of the cortex.
Arterial inflammation | Baseline and 6 months
  Measured as radiotracer uptake in the wall of the thoracic aorta relative to background venous blood uptake via FDG-PET imaging

SECONDARY OUTCOMES:
Heart rate variability | Baseline and 6 months
  Calculated from the average resting heart rate variability collected at baseline and post-treatment visits
Lifestyle factors | Baseline and 6 months
  Self-reported survey results on diet, sleep, and exercise
Earplug use | 6 months
  Time log of earplug use during the study intervention
Stress surveys | Baseline and 6 months
  Self-reported assessments of perceived stress, noise annoyance, and symptoms of depression and anxiety
HOMA-IR | Baseline and 6 months
  Measure of insulin sensitivity performed by blood sample
Leukopoiesis | Baseline and 6 months
  Measured as bone marrow activity via FDG-PET imaging
Blood pressure | Baseline and 6 months
  Systolic and diastolic pressure
MRI based arterial plaque components (such as necrotic tissue and hemorrhage) | Baseline and 6 months
  MRI measurements of atherosclerotic plaque components including necrotic tissue and hemorrhage using black-blood imaging techniques
MRI based arterial wall thickness | Baseline and 6 months
  Measurements of wall thickness as an assessment of atherosclerotic plaque
MRI based brain structure assessments of volume | Baseline and 6 months
  Structural assessment of brain centers to assess volume of neural centers involved in the stress response
MRI based brain connectivity (by measuring changes in blood flow across networks of neural centers at rest and with an emotional task) | Baseline and 6 months
  Connectivity assessment using mapping on functional MRI at baseline and in response to emotional faces of neural centers involved in the stress response to determine the interplay between neural centers before and after therapy by measuring alterations in blood oxygen content under various conditions in different parts of the brain
MRI based brain activation (via measuring blood flow in important neural centers at rest and with an emotional task using functional MRI) | Baseline and 6 months
  Activation assessment using functional MRI at both rest and in response to emotional faces of neural centers involved in the stress response before and after therapy by measuring blood flow under various conditions to different parts of the brain
Axonal integrity of resting neural connections between brain centers using MRI | Baseline and 6 months
  Measurement of axonal integrity using diffusion tensor imaging on MRI to determine the strength connections between important brain centers and neural networks related to stress perception before and after earplugs
MRI based brain structure assessments of density | Baseline and 6 months
  Structural assessment of brain centers to evaluate the density of neural centers involved in the stress response

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osborne, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data necessary for the replication of study results will be made available in deidentified fashion. This includes numerical measurements from imaging, blood tests, and surveys.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the time of manuscript publication or study termination
Access Criteria: These data will be available on an approved data site and will be accessible to the scientific community but will not include any identifying information

REFERENCES:
- [Background] Osborne MT, Radfar A, Hassan MZO, Abohashem S, Oberfeld B, Patrich T, Tung B, Wang Y, Ishai A, Scott JA, Shin LM, Fayad ZA, Koenen KC, Rajagopalan S, Pitman RK, Tawakol A. A neurobiological mechanism linking transportation noise to cardiovascular disease in humans. Eur Heart J. 2020 Feb 1;41(6):772-782. doi: 10.1093/eurheartj/ehz820. PMID 31769799
- [Background] Osborne MT, Naddaf N, Abohashem S, Radfar A, Ghoneem A, Dar T, Wang Y, Patrich T, Oberfeld B, Tung B, Pitman RK, Mehta NN, Shin LM, Lo J, Rajagopalan S, Koenen KC, Grinspoon SK, Fayad ZA, Tawakol A. A neurobiological link between transportation noise exposure and metabolic disease in humans. Psychoneuroendocrinology. 2021 Sep;131:105331. doi: 10.1016/j.psyneuen.2021.105331. Epub 2021 Jun 17. PMID 34183223
- [Background] Sorensen M, Pershagen G, Thacher JD, Lanki T, Wicki B, Roosli M, Vienneau D, Cantuaria ML, Schmidt JH, Aasvang GM, Al-Kindi S, Osborne MT, Wenzel P, Sastre J, Fleming I, Schulz R, Hahad O, Kuntic M, Zielonka J, Sies H, Grune T, Frenis K, Munzel T, Daiber A. Health position paper and redox perspectives - Disease burden by transportation noise. Redox Biol. 2024 Feb;69:102995. doi: 10.1016/j.redox.2023.102995. Epub 2023 Dec 18. PMID 38142584